CLINICAL TRIAL: NCT04215497
Title: Effect of Physiotherapeutic Scoliosis-Specific Exercises on Spine Joint Reposition Sensation in Adolescent Idiopathic Scoliosis
Brief Title: Effect of PSSE on Spine Reposition Sensation in Scoliosis
Acronym: PSSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Zengin Alpozgen, Asst. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/1500
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Scoliosis; Adolescence; Spinal Curvatures; Proprioception; Physiotherapy; Exercise
Keywords: scoliosis; PSSE; proprioception; joint reposition
MeSH Terms: conditions — Scoliosis; Spinal Curvatures; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapeutic Scoliosis-Specific Exercises (Experimental): PSSE group will receive corrective exercise for scoliosis
  Interventions: Other: PSSE
- Control (No Intervention): Control group will be taken to the queue list.

INTERVENTIONS:
Other: PSSE — Physiotherapeutic Scoliosis-Specific Exercises (PSSE) group will receive exercise for 30-40 mins in a day, twice in a week, totally 8 weeks and 16 hours.
  Control group will be taught the basic elements of corrective exercises and want them to do the practising during 8 weeks at home.
  Arms: Physiotherapeutic Scoliosis-Specific Exercises

SUMMARY:
The main aim of the investigator's study is to investigate the effect of Physiotherapeutic Scoliosis-Specific Exercises (PSSE) on spine joint reposition sense and also to investigate the effect of PSSE on vertebral rotation, pain, posture, body image and quality of life in Adolescent Idiopathic Scoliosis (AIS).

Twenty-six patients with AIS will randomly allocated to two groups. 'Schroth' exercises will apply to the PSSE group for 8 weeks (16 sessions). The control group wiil teach basic elements. Patients' spinal pain (Visual Analogue Scale), posture parameters (PostureScreen Mobile, Posterior Trunk Asymmetry Index (POTSI) and Anterior Trunk Asymmetry Index (ATSI)), cosmetic perception (Walter Reed Visual Evaluation Scale (WRVAS)), joint reposition sensations (dual-inclinometer), quality of life (Pediatric Quality of Life Scale and SRS-22) will assess at the first session and at the end of 8 weeks.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional deformity of the spine which is seen in 1-3% of the adolescent population and mostly in girls. Lateral curvature in the frontal plane, axial rotation in the horizontal plane, and kyphosis and lordosis in the sagittal plane are observed. Etiology-related factors of AIS are genetic factors, abnormal neurophysiological functions occurring in the nervous system, hormones, metabolic dysfunction, abnormal skeletal development, biomedical factors, environmental and lifestyle factors.

The vertical position is associated with cortical, subcortical and medullar integration, and postural control based on bodily input.

Approaches as observation, patient education, scoliosis-specific physiotherapy exercises (PSSE), inpatient rehabilitation, electrical stimulation, manipulative applications and brace application are the conservative treatments of scoliosis. PSSE, which includes three-dimensional correction, daily life activities training, posture stabilization and patient education, is a method recommended by Society On Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT) for the conservative treatment of scoliosis. The Schroth 'method is one of the PSSE methods that use three-dimensional postural correction mechanisms. The main goal of the Schroth 'exercises is to reduce the asymmetric load on the spine by using posture variations specific to the patient's curvature. There are no studies i regarding the effect of PSSE on changing proprioceptive neural mechanisms evaluated in the etiopathogenesis of scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* To have diagnosis of Adolescence Idiopathic Scoliosis
* To be in between 10-17 years
* To be the Cobb angle which determined in Anteroposterior graphy as between 10-45 degree
* To not having any other exercise attitude about scoliosis before.
* To attend the programme regularly
* To be volunteer about being participant to the study

Exclusion Criteria:

* Accompanying mental problems, rheumatologic, neuromuscular, cardiovascular, pulmonary history
* The presence of orthopedic problems or pain that prevent to do exercises
* Loss of vision and / or hearing
* Spinal surgery or tumor history
* Diseases in which exercise is contraindicated
* Patients with communication problems

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-25 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of spine joint position reproduction | 8 week
  Acumar™ Dual Inclinometer:
  The subjects will be asked to stay at the reference position for three seconds and then move to the upright position and then go back to the reference angle with their eyes closed. The absolute difference between the two positions in degrees will be noted as the reposition error value. The decrease in the reposition error value is considered as the improvement in the reposition sense.

SECONDARY OUTCOMES:
Spinal pain assessment | 8 week
  Visual Analogue Scale (VAS):
  It is used to quantify the pain intensity of patients. The condition that there is no pain is expressed as 0, and the condition that there is too much pain to be tolerated is expressed as 10.
Frontal-sagittal plan posture evaluation | 8 week
  "PostureScreen Mobile" Application:
  Frontal and sagittal plan posture evaluation will be calculated by marking the reference points on the anterior, posterior and lateral photographs of the patient in "PostureScreen Mobile" application. The total displacement values in the anterior, posterior and lateral directions for postural impairment will be noted in "cm". Decreasing the total displacement values is considered as an improvement in postural parameters.
Body Symmetry | 8 week
  Posterior Trunk Asymmetry Index (POTSI):
  The Posterior Trunk Asymmetry Index parameter is defined as the sum of the six indices: the three frontal plane asymmetry index (C7, axilla folds and waist lines) and the three frontal plane height difference index (acromions, axilla folds and waist lines). The Posterior Trunk Asymmetry Index score is calculated by placing the indices on the posterior photo of the patient. The Posterior Trunk Asymmetry Index score, which represents full symmetry, is '0' and the increase in score indicates increased trunk asymmetry.
Body Symmetry | 8 week
  Anterior Trunk Asymmetry Index (ATSI):
  It is defined as the sum of the six indices determined on the patient's anterior photo: three frontal plane asymmetry indices (stern notch, axilla folds and waist lines) and three frontal plane plane height difference indices (acromions, axilla folds and waist lines). The Anterior Trunk Asymmetry Index score is calculated by placing the indices in the formula. The Anterior Trunk Asymmetry Index score, which represents full symmetry, is '0' and the increase in score indicates increased trunk asymmetry.
Deformity perception assessment | 8 week
  The Walter Reed Visual Assessment Scale (WRVAS):
  It is designed to understand the visual change caused by scoliosis and evaluates deformity under 7 headings. There are 5 different pictures that show different degrees of deformity. Each deformity is scored from 1 to 5; "1" is the best, "5" is the worst. The total score is obtained by summing the scores from all titles and dividing them by 7. The score ranges from 1 to 5, and a higher total score means that the perceived deformity is worse.
Health-related quality of life assessment | 8 week
  Pediatric Quality of Life Inventory:
  This inventory consists of two forms: child and family. Both forms included physical functions (8 items), emotional functions (5 items), social functions (5 items) and school functions (5 items). Scoring is done between 0-5 for each question. The total score of the inventory ranges between 0-100 points. The higher the score represents better the health-related quality of life.
Quality of life assessment for scoliosis: Scoliosis Research Society-22 Questionnaire (SRS-22) | 8 week
  Scoliosis Research Society-22 Questionnaire (SRS-22):
  The questionnaire assesses five domains: function, pain, personal image, mental health (five questions each) and treatment satisfaction (two questions). Each question is scored between 1 (worst) and 5 (best). In the interrogation whose total score ranged from 22 to 111, the high score indicates that the quality of life for scoliosis is better.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Faculty of Health Science, Istanbul, Turkey (Türkiye)